CLINICAL TRIAL: NCT06298409
Title: Evaluating the Effect of Rifaximin on the Regional Composition of the Gut Microbiota and Metabolic Profiles of Subjects With SIBO Using the CapScan® Collection Capsule
Brief Title: Evaluating the Effect Of Rifaximin on the Gut Microbiota and Metabolome in SIBO Using CapScan®
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Envivo Bio Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EB04
Record Dates: First submitted 2024-02-28; First posted 2024-03-07 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Small Intestinal Bacterial Overgrowth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CapScan collection capsule — The CapScan collection capsule is a single-use device that collects fluids from the gastrointestinal tract for analysis ex-vivo.

SUMMARY:
We will sample intestinal microbiota using a microbiome sampling capsule in patients with Small Intestinal Bacterial Overgrowth (SIBO)

DETAILED DESCRIPTION:
Prospective, open-label, single-arm, non-randomized, multi-center study designed to evaluate the effect of the antibiotic rifaximin on the regional composition of the gut microbiota and metabolic profiles of subjects diagnosed with SIBO, using the CapScan collection capsule.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age or older and 80 years of age or younger at the time of the first Screening Visit.
* ASA Classification 1 or 2.
* For women of childbearing potential, negative urine pregnancy test within 7 days of Screening Visit.
* Willingness to use highly effective contraception during the entire study period (e.g.: implants, injectables, oral contraceptives, intra-uterine device or declared abstinence).
* Subject is fluent in English and understands the study protocol and informed consent and is willing and able to comply with study requirements and sign the informed consent form.
* Positive for at least one clinical symptom consistent with SIBO.
* Positive lactulose breath test for SIBO, by Hydrogen (H2) criteria.
* Prescribed, but has not started, a two-week course of Rifaximin for SIBO.

Exclusion Criteria:

* History of any of the following: Prior gastric or esophageal surgery, including lap banding or bariatric surgery, bowel obstruction, gastric outlet obstruction, diverticulitis, inflammatory bowel disease, ileostomy or colostomy, gastric or esophageal cancer, achalasia, esophageal diverticulum, active dysphagia or odynophagia.
* Actively taking a proton-pump-inhibitor medication within 30 days of enrollment
* Pregnancy or planned pregnancy within 30 days from Screening Visit, or breast-feeding
* Any form of active substance abuse or dependence (including drug or alcohol abuse), unstable medical or psychiatric disorder, or any chronic condition susceptible, in the opinion of the investigator, to interfere with the conduct of the study
* A clinical condition that, in the judgment of the investigator, could potentially pose a health risk to the subject while involved in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Sampling of gut microbiota | 56 days
  > 75% of the retrieved CapScan devices to provide at least 3 million metagenomic DNA sequencing reads of gut microbes from the intestinal tract, and at least 900 annotated gut metabolites.
Sampling of gut metabolome | 56 days
  >75% of the retrieved CapScan devices to provide at least 900 annotated gut metabolites.

SECONDARY OUTCOMES:
Effect of rifaximin on gut microbiota | 56 days
  Determine the effect of rifaximin on the regional compositions of the gut microbiota among SIBO patients by assessing the diversity, centroids and distributions of microbial taxa from sequenced CapScan samples of each subject before and after rifaximin at 5 time points.
Effect of rifaximin on gut metabolome | 56 days
  Determine the effect of rifaximin on the regional compositions of the gut metabolites among SIBO patients by assessing the changes to metabolite classes and metabolic pathways as measured by LC/MS-MS analysis of CapScan samples for each subject before and after rifaximin at 5 time points.

CONTACTS AND LOCATIONS:
Overall Officials: George Triadafilopoulos, Principal Investigator — Silicon Valley Gastroenterology
Locations (1):
- Silicon Valley Gastroenterology, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: No